CLINICAL TRIAL: NCT02556008
Title: Cannabidiol for the Treatment of Pediatric Epilepsy (Expanded Access/Compassionate Use Protocol)
Brief Title: Cannabidiol for Pediatric Epilepsy (Compassionate Use)
Status: No longer available | Type: Expanded Access
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Sponsor
Other Study IDs: SH001
Record Dates: First submitted 2015-09-18; First posted 2015-09-22 (Estimated); Last update posted 2026-01-22 (Actual); Status verified 2017-05

CONDITIONS: Refractory Childhood Epilepsy
Keywords: Children; Epilepsy; Cannabidiol
MeSH Terms: conditions — Epilepsy | interventions — Cannabidiol

INTERVENTIONS:
Drug: cannabidiol (CBD) — Treatment will begin with 2 mg/kg/day given in two divided doses. The dose will be increased by 3 mg/kg/day after seven days and then by 5 mg/kg/day every seven days up to a maximum dose of 25 mg/kg/day given.
  Other Names: Epidiolex

SUMMARY:
This is an open-label observational study of pure CBD for the treatment for 25 children with intractable epilepsy. As pure CBD is not FDA approved, the investigators are conducting this study via the FDA expanded access mechanism on a compassionate use basis. The target patient population is children with severe refractory epilepsy who have exhausted all other reasonable avenues of treatment. These are patients for whom the risks of a relatively untested product are outweighed by the potential benefit. Using seizure-diaries maintained on a routine clinical basis, seizure frequency will be assessed four weeks prior to initiation of CBD, one month after CBD initiation, and at least every 3 months thereafter. CBD will be administered as an adjunct to all current anti-epileptic therapies.

DETAILED DESCRIPTION:
Study Overview:

The investigators hope to gain an understanding of the utility of pure CBD use for the treatment of drug resistant epilepsy in this open-label dose-finding observational study. A baseline seizure frequency will be recorded for each subject in a diary for four weeks prior to investigational drug initiation and parents/caregivers will document seizures on a daily basis throughout the study period. Investigational drug (CBD) will be administered as an adjunct to all current anti-epileptic drugs. Once at their maintenance daily dose they will be evaluated one month after achieving the final steady state dose and every three months thereafter.

Visits will consist of neurological exam and seizure diary review. Baseline visit will take 1 hour and each visit thereafter will take approximately 30 minutes.

Safety and Tolerability Measurements:

Data on safety and tolerability of pure CBD is limited. According to the GW Pharma CBD Investigator's Brochure (Appendix G), side effects reported as greater than placebo with highly purified CBD in one clinical trial were conjunctival hemorrhage, change in vision, diarrhea, flatulence, gastric reflux, joint pain, muscle pain, difficulty concentrating, abnormal mood and trouble sleeping.

The patients will be closely monitored for side effects during the titration and treatment period and the dose and/or frequency may be adjusted as appropriate.

CBD is an inhibitor of CYP 2C19, CYP 2C9, and other cytochrome P450s belonging to the 2C and 3A subfamilies. The effects of CBD administered concomitantly with anti-epileptic drugs that are metabolized by this enzyme system are unknown. Anti-epileptic drug doses will be adjusted as needed based on signs and symptoms of toxicity and / or changes in drug levels.

Measurement of changes in seizure frequency:

All seizure types will be classified before study entry. Seizure type and frequency will be monitored during baseline and treatment as recorded in a patient diary. For assessing the efficacy of CBD, the investigator will count only change in the frequency of seizures (ie, tonic seizures, clonic seizures, tonic-clonic seizures lasting more than 3 seconds, atonic seizures, myoclonic seizures including myoclonic absences). In addition, parents/caregivers will report:

* Change in average seizure severity by seizure type, defined as an increase or decrease in seizure duration or intensity
* Change in the number of episodes of status epilepticus, defined as convulsive seizure lasting longer than 10 minutes
* Change in the number of uses of rescue medications
* Change in the number of ER visits/ hospitalizations

Data Safety Monitoring:

The Principal Investigator will review all data relating to safety and tolerability throughout the study, after every third patient has been treated, to monitor study conduct and assess patient safety.

Benefits:

Subject may have a reduction in seizures. This study will help the researchers learn more about the effectiveness and safety of CBD in the treatment of drug-resistant epilepsy. Hopefully this information will help in the treatment of future patients with this condition.

ELIGIBILITY:
Inclusion Criteria:

1. Age criteria between the ages of 1 and 17 years.
2. Documentation of a diagnosis of drug resistant epilepsy as evidenced by failure to control seizures despite appropriate trial of two or more AEDs at therapeutic doses. Documentation must include the diagnosis of epilepsy type or epilepsy syndrome, as well as the underlying cause, when known.
3. Between 1-3 baseline anti-epileptic drugs at stable doses for a minimum of 4 weeks prior to enrollment. Vagus nerve stimulator (VNS), ketogenic diet and modified Atkins diet do not count toward this limit.
4. VNS must be on stable settings for a minimum of 3 months.
5. If on ketogenic diet, must be on stable ratio for a minimum of 3 months
6. Written informed consent obtained from the patient or the patient's legal representative must be obtained prior to beginning treatment.

Exclusion Criteria:

1. Use of any "community acquired" cannabidiol product over the last 3 months.
2. Use of any investigational treatments over the last 3 months.
3. Patients with a history of non-compliance to medical regimens or who are considered potentially unreliable or will not be able to complete entire study.

Ages: 1 Year to 17 Years | Sex: All
Age Groups: Child

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States